CLINICAL TRIAL: NCT00775996
Title: The Objective of This Study Was to Compare the Single-Dose Relative Bioavailability of Ranbaxy and Abbott (Tranxene® T-Tab®) 15 mg Clorazepate Dipotassium Tablets Under Fasting Conditions.
Brief Title: Bioequivalence Study of Clorazepate Dipotassium 15mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA06461
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence Clorazepate Tablets
MeSH Terms: interventions — Clorazepate Dipotassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 15 mg clorazepate dipotassium tablets of ranbaxy
  Interventions: Drug: Clorazepate Dipotassium 15mg Tablets
- 2 (Active Comparator): (TranxeneeT-Tab®) 15 mg clorazepate dipotassium tablets
  Interventions: Drug: Clorazepate Dipotassium 15mg Tablets

INTERVENTIONS:
Drug: Clorazepate Dipotassium 15mg Tablets

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Ranbaxy and Abbott (TranxeneeT-Tab®) 15 mg clorazepate dipotassium tablets under fasting conditions.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioequivalence study on clorazepate dipotassium comparing clorazepate dipotassium 15mg tablets of Ranbaxy Laboratories with Abbott (TranxeneeT-Tab®) 15 mg, in healthy, adult, human, subjects under fasting conditions. A total of 32 subjects, 25 males and 7 females, were enrolled in the study, and 31 subjects, 24 males and 7 females, completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were only included in the study if they met all of the following criteria:

  1. Healthy adult male or female volunteers, 18-55 years of age
  2. Weighing at least 60 kg for males and 52 kg for females and within 15% of their ideal weights
  3. (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983); Medically healthy subjects with clinically normal laboratory profiles and ECGs as deemed by the principal investigator;
  4. Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods:

     * surgically sterile (bilateral ligation, hysterectomy, bilateral oophorectomy) 6 months minimum;
     * IUD in place for at least 3 months;
     * barrier methods (condom, diaphragm) with spermicide from the time of last menstrual period and throughout the study;
     * surgical sterilization of the partner (vasectomy for 6 months minimum);
     * hormonal contraceptives for at least 3 months prior to the first dose of the study. Postmenopausal women with amenorrhea for at least 1 year, and confirmed by blood testing (FSH levels > 40 international units/mL).
* Voluntarily consent to participate in the study,

Exclusion Criteria:

Subjects were excluded from the study if there was evidence of any of the following at screening or at any time during the study:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of:

  * alcoholism or drug abuse;
  * seizures;
  * g1aucoma;
  * hypersensitivity or idiosyncratic reaction to any drug, especially clorazepate or benzodiazepines.
* Female subjects who are pregnant or lactating.
* Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who have made a donation (standard donation amount or more) of blood or blood products (with the exception of plasma as noted below) within 56 days prior to the first dose.
* Subjects who have made a plasma donation within 7 days prior to the first dose.
* Subjects who have participated in another clinical trial within 28 days prior to the first dose.
* Subjects with hemoglobin less than 12_0 g/dL.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2003-08; Primary Completion 2003-09 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html